### HONG KONG BAPTIST UNIVERSITY

### INFORMED CONSENT STATEMENT

[Evaluation of an E-intervention on multiple health behaviour change for Chinese cardiac patients in home-based rehabilitation]

- ---You are invited to participate in a research study. The purpose of this study is to provide you an innovative and comprehensive intervention program targeting rehabilitation exercise and dietary behaviour, which you can follow at home after you discharge from rehabilitation in hospital. The outcomes of this research project will provide knowledge relative to:
- 1. Examining whether participants in the intervention program increase their physical activity (PA) levels and fruit and vegetable intake (FVI) portion compared to the control group.
- 2. Examining whether the intervention program can improve participants' social-cognitive variables of PA and FVI.
- 3. Examining whether the intervention program can improve participants' perceived quality of life and decrease depression level.

## **INFORMATION**

Before you participate in this study, please first check whether you meet the following inclusion criteria or not. (1) Participants should be 18 years old or above; (2) no restriction of physical mobility under the cardiac function at entry; and (3) no restriction of relevant disease such as diabetes or fruit allergies.

If you meet above criteria and are willing to participate in this study, you will receive an eight-week online intervention after you discharge from rehabilitation. You are required to access to an e-health website once per week during this program period. Each elearning session will cost approximately 15 minutes in average. The internet website contains several learning modules, such as information pages regarding how to engage in appropriate physical activity and maintain healthy dietary, digital personalized agenda in which you formulate your activity plans, nutrition plans, as well as health model learning to increase your motivation and self-confidence on physical activity and nutrition. During the intervention, you will also simultaneously receive a SMS message via mobile phone each week reminding you to access your weekly session. Besides, you will be further contacted for collecting data at the beginning of intervention (T1), at the end of intervention (T2), and 1 month after the intervention (T3). Each electronic questionnaire survey will last approximately 15 minutes. All website hyperlinks for the questionnaire surveys at T1, T2, and T3 as well as for the weekly e-health learning session will be delivered by Wechat of mobile phone.

All information you provided will be kept strictly confidential. Only the results of statistical analyses will be reported. Please indicate your true perception or feeling about issues described in the questionnaire.

## **RISKS**

There is no any potential risk or discomforts related to the intervention conduction.

## **BENEFITS**

After you discharge from rehabilitation in hospital, you will obtain supporting information about physical activity and dietary behaviour by the way of e-health learning at home, in the long-term, which might not only maintain the intention, increase planning, coping abilities and well-being, but might also facilitate the return to work process.

## CONFIDENTIALITY

We will collect your data via study website, which is built by us. One category of data is your personal information including name, gender, age, mobile phone No., place of residence, marital status, number of children, education level, current work status etc. However, as the data is on the internet, we cannot guarantee confidentiality.

The identifiers will be destroyed within 3 years upon completion of our research study.

## **COMPENSATION**

You will receive cash <u>RMB 50</u> once the completion of intervention and online questionnaires survey across three measurement time points. If you withdraw from the study prior to its completion, you won't receive it.

## **CONTACT**

If you have questions at any time about the study or the procedures, you may contact the researcher, <u>Dr. Duan Yanping</u> at <u>852-34113080</u> or <u>duanyp@hkbu.edu.hk</u>. The address is <u>Hong Kong Baptist University Shek Mun Campus, 12/F, 8 On Muk Street, Shek Mun, Shatin, Hong Kong.</u> If you feel you have not been treated according to the descriptions in this form, or your rights as a participant in research have been violated during the course of this project, you may contact the Committee on the Use of Human 7 June, 2018

| and Animal Subjects in Teaching and Research by | email at hasc@hkbu.edu.hk | or by mail to Graduate | School, Hong Kong Baptist |
|---|---|---|---|
| University, Kowloon Tong, Hong Kong | | | |

| | | | _ |
|-------|-------|--------|-----|
| Subje | ect's | initia | als |

## **PARTICIPATION**

Your participation in this study is voluntary; you may decline to participate without penalty. If you decide to participate, you may withdraw from the study at any time without penalty and without loss of benefits to which you are otherwise entitled. If you withdraw from the study before data collection is completed your data will be returned to you or destroyed.

# **CONSENT**

| I have read and understand the above information. I have received a copy of this form. I agree to participate in this study. | |
|---|---|
| Signature of the Subject | Date |
| Signature of the Investigator | Date |

Hong Kong Baptist University 7 June, 2018

7 June, 2018